CLINICAL TRIAL: NCT02423369
Title: Cerebral Oxymetry and Neuronal Biomarkers in Newborns and Infants During Perioperative Period
Brief Title: Cerebral Oxymetry and Neuronal Markers in Newborns and Infants Undergoing Surgery
Acronym: NEMARKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Research Council of Lithuania (Other)
Responsible Party: Principal Investigator, Danguole C Rugyte, MD, PhD., Lithuanian University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BE-2-43
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Peri-operative Injury; Newborn, Infant, Disease
Keywords: S-100B protein; Neuron-specific Enolase
MeSH Terms: conditions — Disease | interventions — S100 Calcium Binding Protein beta Subunit; Blood Specimen Collection; Phosphopyruvate Hydratase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neonates and infants requiring surgery (Experimental): neonates and infants in whom blood samples for measurement of S-100 B protein in serum and NSE protein in serum are taken pre-operatively and 1-st, 2-nd and 3-rd post-operatively. During anesthesia cerebral near infrared spectroscopy is continuously applied until the wound closure.
  Interventions: Procedure: Cerebral near infrared spectroscopy; Other: S-100B protein in serum; Other: NSE protein in serum

INTERVENTIONS:
Procedure: Cerebral near infrared spectroscopy — At the start of anesthesia on the patient's forehead two electrodes are attached the for continuous measurement of cerebral near infrared spectroscopy during surgery.
  Other Names: cerebral tissue oxygen saturation; cerebral oxymetry
Other: S-100B protein in serum — 0,5-1 ml of blood from periferal site for determination of serum S-100B concentration.
  Other Names: S-100B protein in blood
Other: NSE protein in serum — 0,5-1 ml of blood from periferal site for determination of serum NSE concentration.
  Other Names: Neuron-specific Enolase in blood

SUMMARY:
The purpose of this study is to assess whether peri-operative period in neonates and infants is associated with an increase in blood biomarkers, specific for neuronal injury, and to correlate them with clinical variables and sedative/analgesic agents. Patients, who meet inclusion criteria and does not meet exclusion criteria, are enrolled. Blood samples for measurement serum concentrations of markers (S100-B and Neuron-Specific Enolase (NSE)) are drawn before surgery (baseline) and on the 1-st, 2-nd and 3-rd day after surgery. During surgery cerebral oxygenation (rSO2) monitoring is continuously applied; rSO2, hemodynamic and respiratory values are simultaneously recorded every 5 minutes. Anesthesia, pre and postoperative treatment, including analgesia and sedation, are given as per standard of care.

DETAILED DESCRIPTION:
Retrospective studies have shown that surgery in infancy is associated with worse neurodevelopmental outcome, compared to general population. The reasons may be complex, and patients at risk are unknown. Brain growth and central nervous system formation are extremely active in neonates and infants. Metabolic or circulatory derangement may have negative influence on the developing brain. Disease and perioperative period, both may further put this population at risk for physiological abnormalities. Near infrared spectroscopy was shown to be a convenient method for monitoring of cerebral tissue oxygenation during surgery.

The great majority of anesthetics and sedative drugs, used in perioperative period, were shown to cause neuronal apoptosis in experimental animals. Some studies found that neurological marker S-100B increased in cerebrospinal fluid and blood immediately following anesthesia in animals. Several clinical studies supported this founding in children following cardiac and general surgery.

The aim of this study is to assess the dynamics of S-100B protein pre- and during 72 hours after surgery in neonates and infants aged 1-93 days, operated for abdominal/thoracic/urologic malformations/disease. As S-100B in blood may have extracranial sources, we simultaneously assess other neuronal marker Neuron-specific Enolase.

ELIGIBILITY:
Inclusion Criteria:

* patients, undergoing general, thoracic, urological surgery for congenital anomalies or disease
* signed written informed consent by parents/official caregivers

Exclusion Criteria:

* cardiac surgery
* any evidence of neurological disease
* sepsis
* limited ability to obtain blood samples
* clinically significant anemia
* physical status of the patients corresponding to American Society of Anesthesiologists (ASA) class 4 and 5.

Max Age: 93 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
change in S-100B and NSE concentrations in serum | within 24 hours and 3 days after surgery
  change in S-100B and NSE concentrations in serum compared to preoperative value

SECONDARY OUTCOMES:
association of S-100B and NSE concentrations in serum with intraoperative cerebral near infrared spectroscopy values. | within 24 hours after surgery

OTHER OUTCOMES:
association of S-100B and NSE concentrations in serum with cumulative doses of sedative agents | within 24 hours pre surgery to 3 days after surgery
  Pre and postoperative S-100B and NSE concentrations in serum will be correlated with the administered pre and postoperative cumulative doses of sedatives and analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Danguole C Rugyte, MD. PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania

REFERENCES:
- [Background] Wang S, Peretich K, Zhao Y, Liang G, Meng Q, Wei H. Anesthesia-induced neurodegeneration in fetal rat brains. Pediatr Res. 2009 Oct;66(4):435-40. doi: 10.1203/PDR.0b013e3181b3381b. PMID 20016413
- [Background] Robertson DR, Justo RN, Burke CJ, Pohlner PG, Graham PL, Colditz PB. Perioperative predictors of developmental outcome following cardiac surgery in infancy. Cardiol Young. 2004 Aug;14(4):389-95. doi: 10.1017/S104795110400407X. PMID 15680045
- [Background] Tina LG, Frigiola A, Abella R, Tagliabue P, Ventura L, Paterlini G, Li Volti G, Pinzauti S, Florio P, Bellissima V, Minetti C, Gazzolo D. S100B protein and near infrared spectroscopy in preterm and term newborns. Front Biosci (Elite Ed). 2010 Jan 1;2(1):159-64. doi: 10.2741/e78. PMID 20036866
- [Background] Vicente E, Tramontina F, Leite MC, Nardin P, Silva M, Karkow AR, Adolf R, Lucion AB, Netto CA, Gottfried C, Goncalves CA. S100B levels in the cerebrospinal fluid of rats are sex and anaesthetic dependent. Clin Exp Pharmacol Physiol. 2007 Nov;34(11):1126-30. doi: 10.1111/j.1440-1681.2007.04687.x. PMID 17880365
- [Background] Jensen E, Sandstrom K, Andreasson S, Nilsson K, Berggren H, Larsson LE. Increased levels of S-100 protein after cardiac surgery with cardiopulmonary bypass and general surgery in children. Paediatr Anaesth. 2000;10(3):297-302. doi: 10.1046/j.1460-9592.2000.00522.x. PMID 10792747
- [Derived] Razlevice I, Rugyte DC, Strumylaite L, Macas A. Assessment of risk factors for cerebral oxygen desaturation during neonatal and infant general anesthesia: an observational, prospective study. BMC Anesthesiol. 2016 Oct 28;16(1):107. doi: 10.1186/s12871-016-0274-2. PMID 27793105